CLINICAL TRIAL: NCT00687830
Title: A Randomized Endoscopist-blinded Clinical Trial Comparing the Bowel Cleansing Effect and Patient Tolerability of Same Day Polyethylene Glycol Bowel Preparation Regimen v Regimen Given on the Day Before Colonoscopy
Brief Title: Efficacy of Morning-only Bowel Preparation for Afternoon Colonoscopy.
Acronym: CCF
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Cleveland Clinic Florida (Other)
Responsible Party: Sponsor
Organization: The Cleveland Clinic (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: CCFL-8964
Record Dates: First submitted 2008-05-28; First posted 2008-06-02 (Estimated); Results first posted 2016-04-11 (Estimated); Last update posted 2017-05-17 (Actual); Status verified 2016-02

CONDITIONS: Colon Cancer
Keywords: Afternoon colonoscopy; Morning; Evening; Bowel Preparation; Efficacy; Satisfaction
MeSH Terms: conditions — Colonic Neoplasms; Personal Satisfaction | interventions — Golytely

STUDY DESIGN:
Who Masked: Care Provider
Oversight: Data Monitoring Committee: No

ARMS (2):
- Polythylene Glycol (PEG) in the evening (Active Comparator): Bowel preparation with Polyethylene Glycol given in the evening prior to the day of the afternoon colonoscopy.
  'Polyethylene Glycol afternoon'
  Interventions: Drug: Polyethylene Glycol afternoon
- Polythylene Glycol (PEG) in the Morning (Experimental): Bowel preparation with Polyethylene Glycol given on the morning of the day of the afternoon colonoscopy.
  'Polyethylene Glycol morning'
  Interventions: Drug: Polyethylene Glycol morning

INTERVENTIONS:
Drug: Polyethylene Glycol afternoon — Prescribed the standard dose of 4L or 1 Gallon Polythylene Glycol to be taken over a period of 4 hours with water. For Evening prep, between 5PM and 9PM
  Other Names: GoLytely
  Arms: Polythylene Glycol (PEG) in the evening
Drug: Polyethylene Glycol morning — Prescribed the standard dose of 4L or 1 Gallon Polythylene Glycol to be taken over a period of 4 hours with water. For Morning prep, between 6AM and 10AM
  Other Names: Golytely
  Arms: Polythylene Glycol (PEG) in the Morning

SUMMARY:
The study aims to study the adequacy of bowel preparation (colon cleansing) for afternoon colonoscopies. The conventional regimen of giving bowel prep on the evening prior to the day of the colonoscopy will be compared with that given on the morning of an afternoon colonoscopy. Endoscopist scoring the bowel cleansing efficacy with an Ottawa Scale are blinded to the randomization process.

DETAILED DESCRIPTION:
Two bowel preparation regimens of Polyethylene Glycol (PEG), commonly referred to as "Golytely" will be tested for their efficacy (bowel cleansing effect) and patient tolerability. The goal is to reduce the failure rates of afternoon colonoscopies, for which, one of the main reasons attributed is inadequate bowel preparation. For the afternoon colonoscopies, the conventional PEG regimen given on the evening prior to the day of the colonoscopy will be compared with the novel PEG regimen given on the morning of the day of the colonoscopy. The comparison will be drawn for two measures - bowel cleansing effect measured from the questionnaire given to the gastroenterologists performing the colonoscopy and the patient tolerability evaluated from the information gathered from the patient's questionnaire.

ELIGIBILITY:
Inclusion Criteria:

* All patients attending the GI Clinic at CCF who are prescribed colonoscopy and are willing to get the procedure done in the afternoon.

Exclusion Criteria:

* Colonoscopy is contraindicated
* Prior Colectomy or colon surgery.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 136 (Actual)
Dates: Start 2008-02; Primary Completion 2009-07 (Actual); Study Completion 2009-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Shibu Varughese, M.D., Principal Investigator — Cleveland Clinic Florida
Locations (1):
- Cleveland Clinic Florida, Weston, Florida, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Varughese S, Kumar AR, George A, Castro FJ. Morning-only one-gallon polyethylene glycol improves bowel cleansing for afternoon colonoscopies: a randomized endoscopist-blinded prospective study. Am J Gastroenterol. 2010 Nov;105(11):2368-74. doi: 10.1038/ajg.2010.271. Epub 2010 Jul 6. PMID 20606677
- See also: European society of GI endoscopy guidelines on bowel preparation. Reference 61, Page 145 : Same day regimen. — http://www.esge.com/assets/downloads/pdfs/guidelines/2013_bowel_preparation_for_colonoscopy.pdf

RESULTS

PARTICIPANT FLOW:
Groups:
- Evening: Bowel prep given in the evening prior to the day of the afternoon colonoscopy
- Morning: Bowel prep given on the morning of the day of the afternoon colonoscopy
Period: Overall Study
Arm/Group | Evening | Morning
Started | 68 | 68
Completed | 68 | 68
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Evening | Morning | Total
Number analyzed (Participants) | 68 | 68 | 136
Age, Continuous [Mean (Standard Deviation); unit: years] | 52.2 (11.5) | 51.4 (10.2) | 51.8 (10.8)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 30 | 35 | 65
  Male | 38 | 33 | 71

OUTCOME MEASURES:

1. Primary Outcome: Comparing All Morning Bowel Prep to Evening Bowel Prep for Patients Undergoing Afternoon Colonoscopies. (Using Ottawa Scale Scores, Range 0-14) Lower Score Indicates a Better Outcome.
Time Frame: Within 1 hr after the colonoscopy procedure
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Evening | Morning
Number analyzed (Participants) | 68 | 68
units on a scale | 7.1 (2.7) | 4.7 (2.4)
Statistical Analysis 1: Comparison: Evening vs Morning; Test type: Superiority or Other; p < 0.01, t-test, 2 sided

2. Secondary Outcome: Patient Satisfaction in the Two Groups, All Morning Prep vs. All Evening Bowel Prep.
Description: Variable used to assess patient satisfaction: Loss of sleep. The numbers below depict the number of participants who experienced loss of sleep.
Time Frame: An hour before the colonoscopy procedure
Measure: Number; unit: participants
Arm/Group | Evening | Morning
Number analyzed (Participants) | 68 | 68
participants | 21 | 11
Statistical Analysis 1: Comparison: Evening vs Morning; Test type: Superiority or Other; p = 0.04, Chi-squared

ADVERSE EVENTS:
Arm/Group | Evening | Morning
Serious Adverse Events (participants affected / at risk) | 0/68 | 0/68
Other Adverse Events (participants affected / at risk) | 0/68 | 0/68

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes